CLINICAL TRIAL: NCT00674063
Title: A Randomized, Double-Blind, Multicenter Study Comparing the Efficacy and Safety of Weekly Intravenous Administration of 7.5mg and 0.075mg/kg Alefacept in Subjects Weighing Between 100kg and 150kg, With Moderate to Severe Chronic Plaque Psoriasis
Brief Title: A Study to Assess the Efficacy and Safety of Two Dosing Regimens of Alefacept in Subjects Weighing Between 100kg and 150kg With Moderate to Severe Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C-738
Record Dates: First submitted 2008-05-06; First posted 2008-05-07 (Estimated); Last update posted 2014-08-26 (Estimated); Status verified 2014-08

CONDITIONS: Chronic Plaque Psoriasis
Keywords: Chronic Plaque Psoriasis; Alefacept
MeSH Terms: interventions — Alefacept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Dose regimen 1
  Interventions: Drug: alefacept
- 2 (Experimental): Dose regimen 2
  Interventions: Drug: alefacept

INTERVENTIONS:
Drug: alefacept — IV
  Other Names: Amevive; ASP0485

SUMMARY:
Comparison of two dosing regimens of Alefacept in subjects weighing between 100kg and 150kg with moderate to severe Chronic Plaque Psoriasis

ELIGIBILITY:
Inclusion Criteria:

* Body weight between 100kg and 150kg
* Diagnosis of Chronic Plaque Psoriasis with Body Surface Area (BSA) involvement of ≥ 10%
* Candidate for phototherapy or systemic therapy for Psoriasis
* CD4 + T lymphocyte counts > lower limit of normal

Exclusion Criteria:

* Clinically significant abnormal hematology values or blood chemistry values
* ALT or AST value of ≥ 3x the upper limit of normal
* Other types of Psoriasis
* Serious infection within 3 months prior to 1st dose of study drug
* Antibody positive for HIV
* History of malignancy
* History of severe allergic or anaphylactic reactions
* History of any clinically significant cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal and/or other major disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2003-07; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects receiving a Psoriasis Area and Severity Index (PASI) score of ≥75 compared to baseline | 1 Week post treatment

SECONDARY OUTCOMES:
Proportion of subjects in each dosing regimen receiving a PASI score of ≥75 compared to baseline | 1 Week post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Use central contact, Study Director — Astellas Pharma US, Inc.
Locations (17):
- United States (11):
  - Hot Springs, Arkansas
  - Fridley, Minnesota
  - Omaha, Nebraska
  - East Windsor, New Jersey
  - Stony Brook, New York
  - Lake Oswego, Oregon
  - Portland, Oregon
  - Johnston, Rhode Island
  - Goodlettsville, Tennessee
  - Nashville, Tennessee
  - Norfolk, Virginia
- Canada (6):
  - Moncton, New Brunswick
  - Hamilton, Ontario
  - London, Ontario
  - Waterloo, Ontario
  - Windsor, Ontario
  - Montreal, Quebec